CLINICAL TRIAL: NCT07399106
Title: EN-CAMHS 2: Enhancing CAMHS Referrals
Brief Title: Enhancing Child and Adolescent Mental Health Service Referrals 2
Acronym: EN-CAMHS 2
Status: Not yet recruiting | Type: Observational
Sponsor: Greater Manchester Mental Health NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Principal Investigator, Kathryn Abel, Professor Kathryn M Abel, University of Manchester
Other Study IDs: GreaterManchesterMentalHealth; NIHR158809 (Other Grant/Funding Number: National Institute for Health and Care Research UK)
Record Dates: First submitted 2025-08-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: No Conditions; Improving Referrals Into NHS CAMHS
Keywords: CAMHS; mental health; digital mental health; referral; stakeholder consultation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Work Package 1 — Requirements Prioritisation
  We shall hold 2 x roundtable events (Manchester and London) to gather feedback and input from senior stakeholders (e.g. NHS England senior leaders; commissioners, CAMHS leaders).
  With our partner MQ, we shall conduct 6 stakeholder focus groups with CYP, families/carers and professionals including GPs, to collaboratively prioritise requirements (identified in EN-CAMHS 1) for the revised digital tool. We aim to recruit up to 10 stakeholders per group, therefore 60 participants in total. We shall use the MoSCoW prioritisation method [29] collaboratively as we have done in a number of other NIHR funded digital health projects. As part of this prioritisation process, each of the existing 11 interactive CAMHS referral forms created by individual CAMHS in England will be rated using the System Usability Scale [30] and using criteria from the EN-CAMHS 1 focus groups e.g. navigability, clarity of language, accessibility.
Other: Work Package 2 — Co-Design and Tool Implementation
  Onboard 5-8 CAMHS providers (with different characteristics and served populations) who are willing and can support an evaluation of the digitally-enhanced CAMHS tool in collaboration with our partners, NHS England.
  Workshops with 5-8 Trust staff from each provider. Co-design the tool with CAMHS stakeholders (2 x 1-hour workshops with 25 referrers).
  Ensure accessibility support (WCAG2.2 and assistive technology, translations of the tools etc) is extensive and supports needs identified by stakeholder consultation (Digital Accessibility Working Group n=10) and in collaboration with PPIE, YPAG and PPAG. This group will be formed from the project with characteristics derived from accessibility needs identified in the stakeholder codesign groups and from ENCAMHS 1. This group shall meet twice during the co-design process to review the tool and suggest accessibility enhancements. Every effort will be made to incorporate suggestions made by this group.
Other: Work Package 3 — Evaluation of Implementation
  Evaluate implementation of the new digitally-enhanced referral process with 60 key referrers.
  Explore the potential, enablers and barriers of embedding a new CAMHS referral mechanism via semi-structured qualitative interviews with 25 referrers.
  Develop a blueprint and toolkit for CAMHS to implement the referral tool. Understand if and how the tool enhances the CAMHS referral process.
Other: Work Package 4 — The charity MQ Mental Health Research was a key partner to EN-CAMHS 1. We plan to continue this successful partnership in EN-CAMHS 2. In this WP4, MQ will drive the sustainability of the EN-CAMHS tools. MQ are actively engaged in discussions with the Prudence Trust about longer-term sustainability support for the platform. MQ aim to collaborate to drive and support the tools' implementation, nationally if possible. This will require lobbying key national stakeholders (including senior policymakers, regional ICB leads, mental health professional bodies) to support implementation of the platform for the medium and longer terms, beyond the lifetime of this grant. MQ have secured funding from the Prudence Trust to support longer term sustainability for the referral tool and enhanced referral processes developed through this project.

SUMMARY:
Background

Increasing numbers of children and young people are being referred to Child and Adolescent Mental Health Services (CAMHS). However, a quarter are 'rejected' for treatment. This can happen for simple reasons like:

1. confusion about what support CAMHS can and cannot provide
2. lack of information about available non-CAMHS support
3. the paperwork submitted to CAMHS is incomplete Being rejected by CAMHS is distressing for children and young people and families. The current process also costs the NHS because of wasted clinical time reviewing children and young people who do not need CAMHS' help. For GPs and school staff making referrals, rejection is frustrating especially if no other help is offered. In the previous NIHR-funded ENCAMHS 1; project, the project team spoke to many children and young people and families with experience of trying to get help from CAMHS. The project team asked the stakeholders about the problems they had and what solutions might help.

Aims This project aims to develop a simple, clear way for children and young people to get the right support for their mental health problems when they need it. This project aims to solve the problems people told us about and to improve the quality of referrals made to CAMHS.

Design & Methods

The project team shall:

* work with all relevant groups including children and young people and families to build a better referral process
* make an easy-to-use digital referral process for CAMHS
* make everything built useful and easy to use for as many people as possible
* provide GPs, school staff and parents with information about non-CAMHS support
* learn how to embed the new referral system across NHS systems (e.g. NHS app)
* test the new process across 5-8 different CAMHS e.g. in and outside cities
* ask people who tested the new process if they liked it and found it useful
* analyse information collected to see how people used it
* work with the charity MQ to make sure what is built is used widely

The project team shall talk to children and young people, families, GPs, school staff, CAMHS staff and policymakers and build the new referral process with the project team. The project team shall hold several workshops which will shape the new digital tools, and ensure the project team considers how to include the right non-digital supports. The project team shall test the new process across 5-8 CAMHS and use a mix of statistical and interview data to understand if the new referral process is valued, useful and easy to use. The project team's partner, MQ, will develop a plan to roll out the tool nationally and to support its use in the long term.

Patient & Public Involvement The project team shall build on established collaborations with young people, their parents/carers/families. The project teamwon a national award for public involvement in the ENCAMHS 1 project. The project team shall be advised throughout by the Young People's Advisory Group (YPAG) and by the Parents and Professionals Advisory group (PPAG). The YPAG and PPAG from the ENCAMHS 1 project have told the project team they would like to work with the project team again on this project. The project team shall also recruit new members.

Dissemination The project team want this project to transform how children and young people get access to appropriate mental health support and to reduce some of the pressures on CAMHS. The project team shall share learning with national NHS bodies. The project team shall make the digital tools the project team builds widely available through the networks. The project team shall publish the academic findings and share widely through social media and mental health partner networks.

DETAILED DESCRIPTION:
BACKGROUND Children and young people's mental health is a national priority for the Department of Health and Social Care [1] and all major national funders. This research addresses critical problems in the referral processes to Child and Adolescent Mental Health Services (CAMHS) that the project team identified during the project team's qualitative research program during the project team's NIHR HS&DR-funded EN-CAMHS 1 project.

1. CAMHS cannot cope with the growing numbers of referrals. Nearly 500,000 children and young people (CYP) were referred to CAMHS in 2021/2022 [2], and this number has risen steadily since 1999 [3,4]. CAMHS providers are overwhelmed by the number of referrals [5,6].
2. Rising demand is coupled with high levels of rejection. Almost a quarter of the referrals made into CAMHS are unsuccessful because they are deemed inappropriate or do not reach the threshold for treatment [2]. This results in longer delays for children who need the specialist care, which is exacerbating mental health difficulties [7].
3. The experience of the referral process is poor [8,9]. The high rate of inappropriate referrals causes unnecessary distress to children, their families and to referrers, who can wait many weeks if not months for a decision [10]. The family upset is compounded by a lack of communication throughout the long process [11]. When a referral is rejected, it typically goes to the 'back of the queue', resulting in further delays for children and families.
4. The quality of CAMHS referrals is poor and CAMHS is often seen as the gold standard by families or the only alternative by referrers struggling to know what else is available in primary care [7,10].
5. Clear information about what CAMHS can and cannot provide is not readily available and suitable alternative sources of mental health support are often not explained to children and their families at the point of referral rejection [12,13].
6. Non-CAMHS support is poorly understood [14] and not widely valued as a helpful source of support. People who could be helped better by non-CAMHS support are not signposted elsewhere early enough in the process, except in a minority of places.
7. Rejected referrals incur a significant cost for CAMHS who must triage often incomplete and/or inaccurate, referral documentation. Receiving a rejection is also frustrating and costly to referrers (GPs, school staff) who spend valuable time preparing referral documentation [15,16].

The NIHR funded EN-CAMHS project ("EN-CAMHS 1", NIHR131379) consulted with 110 CAMHS stakeholders (CYP, parents/carers, GPs, mental health school staff and CAMHS professionals) [17]. EN-CAMHS 1 confirmed and extended previous research: stakeholders reported widespread confusion about the kinds of support CAMHS can and cannot provide. Referrers reported poor support during the referral process, lack of transparency about the process and a lack of knowledge and low confidence in other sources of support. Services reported poor quality of referrals such that many were 'rejected'. Families described using 'workarounds' to get to CAMHS (e.g. going to A&E). This is concerning not least because it highlights families' difficulties, but also because it disrupts the goals of referral and triage: i.e. to provide timely, appropriate care and to prioritise those in most need. The project team identified overwhelming problems with the current referral processes resulting in high levels of unnecessary additional cost to services; and widespread despair for referrers and for children and families.

RATIONALE Direct changes to CAMHS resourcing and staffing are the domain of DHSC and not something the project team can change. However, by improving referrals, the work can relieve additional pressure on services, make the process work better and create greater satisfaction for users. The project team can also increase understanding of what CAMHS is and does; and create confidence in CAMHS alternatives. The research has demonstrated an urgent health and care need to provide a straightforward referral process to ensure that children most in need are prioritised for treatment, and that all children are signposted to appropriate help in a timely manner. Such a process needs to be scalable, low cost, widely accessible and sustainable over time.

110 CAMHS stakeholders in EN-CAMHS 1 [18] repeatedly expressed a clear preference for a digital solution that could simplify and improve the CAMHS referral process. Stakeholders unanimously advised that the project team should create a national, standardised referral process which could also be tailored to local CAMHS' configurations. To date, there has been no national collaboration to improve the referral process; rather, piecemeal attempts across CAMHS providers have adopted different approaches. The project team's audit of such approaches unfortunately suggests referrals do not meet the requirements of CAMHS stakeholders identified in EN-CAMHS 1. For example, none has been rigorously co-developed with stakeholders; none provides a mechanism for people to track 'where they are' in the referral journey once a referral is submitted. From a technical perspective, the digital tools currently developed are not interoperable with core NHS infrastructure (e.g. NHS app; NHS website). There is patchy sharing of digital referrals in geographically-aligned providers, but it is fragmented and again lacks most of the recommendations the project team brings from EN-CAMHS 1 stakeholders for what the digital referral should 'look like'.

EN-CAMHS 1 stakeholders recommended the project team implement a digital solution to address the current problems of poor communication, missing information, poor data quality and lack of guidance for families about what to expect of the referral journey. The design and development of the digital tool will specifically address the accessibility needs of referrers. The project team intend to explore issues of digital accessibility in the consultations (WP1) and in the co-design workshops with participants. The project team shall also consider the three key elements of digital exclusion: lack of digital access; lack of digital skills; lack of confidence to use digital. The project team will explore these challenges in the co-design workshops, with stakeholders in consultation and with advisory groups. The digital tool will supplement rather than supplant traditional modes of referral; traditional (e.g. paper based) modes of referral will remain. However, the project team anticipates that the project team's digital tool will enable more people to make more successful referrals than before.

The project team shall also generate new knowledge about the patterns of referrals into CAMHS, by automating data collection through the digital tools and thereby enabling services and NHS England to understand referral and treatment data in greater detail than ever before. The project team see enormous potential in this project and its learnings/outputs for cross-pollination to other services experiencing similar problems.

1. Referrals overwhelming CAMHS The project team cannot increase CAMHS staff levels or change what it can provide.

   The project team can make the referral process work better and with greater satisfaction for referrers and for those being referred.

   The project team can increase confidence in CAMHS alternatives and increase follow-through into CAMHS alternatives.

   The project team can help CAMHS prioritise the needs of those it is designed to help.
2. Quality of referrals is poor The project team can provide clear, accessible guidelines to make appropriate referrals.

   The project team can validate input on the referral form and ensure all required information is completed pre-submission.

   The project team can raise awareness about what a good referral is. The project team can educate people about common referral mistakes.
3. Poor experience of referral The project team can explain the referral process clearly. The project team can outline key steps in the referral journey and inform people about the expected waiting times for the local CAMHS triage process.

   The project team can update referrers and CYP/families as their referral moves through the system.

   The project team can signpost to local and national resources that may help during the waiting period.
4. Costs for CAMHS The project team can reduce CAMHS clinical time wasted by automating the checking of referral documents before they are submitted.

   The project team can reduce costs for individual and families by streamlining this process.

   The project team can improve referral success by ensuring alternative non-CAMHS support is signposted appropriately and explained.
5. Poor information The project team can provide straightforward accessible information translated into multiple languages.

   The project team can signpost to phoneline support for those who are not comfortable with technology.
6. Lack of confidence in non-CAMHS The project team can make non-CAMHS support more understandable and transparent to people using services by linking to real-life case studies / CYP stories and working with CAMHS stakeholders.

   The project team can help build trust between referrers and services.
7. Timeliness of Assessment by CAMHS The project team can divert CYP to alternative services which may free CAMHS to see those who need CAMHS most, sooner.

The project team can reduce the workload of CAMHS staff in triaging inappropriate referrals.

The project team can free up CAMHS clinical time for more complex appropriate referrals.

The project team can make referrals faster and more reliable. The project team can make referrals 'recyclable' so re-referrals do not 'fall out' of the system and need to 'start from scratch'/'go back to the back of the queue.'

EVIDENCE The number of children and young people (CYP) waiting longer than 12-weeks for mental health treatment in England is at a five-year high [19]. The challenge for CAMHS improvement is complex, but a review of the current literature has identified how the referral process represents an important aspect of this leading to children waiting until they are very unwell to access care [10,19]; possibly needing more prolonged and intensive treatment as a result and leading to lack of trust in services [20,21]. Simple, practical problems already identified in the literature include lack of transparency in the referral process; incomplete information in referral forms; poor communication with referrers/families throughout the process; lack of information about where else to seek help and who can refer into CAMHS [e.g. 22-25]. The NIHR HS&DR-funded EN-CAMHS 1 extended this understanding of the challenges for referrals into CAMHS.

Existing evidence suggests potential solutions include: a 'single point of access' (SPoA) within CAMHS [e.g. 26-28] referrer-friendly guidelines with training to support referrers [14]; increasing, and ring-fencing funding available to CAMHS [6]; clarity about CYP mental health support available for referrers that is separate from CAMHS and which may be more readily and repeatedly available in the community [9,27]; and a call for policymakers to improve collaboration between professionals involved in supporting CYP mental health [11]. However, an audit of CAMHS referral processes found that only 11 providers (out of 78) have online, interactive referral forms, many of which have poor user interfaces and are difficult to navigate. Most have no online referral mechanism and provide lengthy documents that need to be downloaded, printed and/or emailed individually to each different provider. Referrers told the project team these forms were often hard to find, confusing and difficult to complete. Easy-win opportunities to provide online referral forms that automatically validate information and support accessibility (e.g. translations) have not been exploited. Other helpful information, such as: overviews of what CAMHS can and cannot provide, indicative waiting times, signposting to alternative local sources of help and other support mechanisms are not available in a standardised format. Children and families told the project team they did not know where to find information about CAMHS and that they did not know which sources of information to trust. Opportunities for co-designed, patient-centred communications accessible to this (and other) marginalised and under-represented groups have been missed.

EN-CAMHS 1 engaged widely with children and families, policymakers, commissioners, mental health staff, NHS England and other CAMHS stakeholders to identify the key problems and the tractable solutions to the CAMHS referral problems. Stakeholders advocated for a digitally-led referral process that would support completeness of submitted information; signpost to alternative help and resources (where applicable); real-time updates about where a child is on the referral pathway and approximate waiting times to referral outcomes and treatment. Mental health staff identified time-savings that would accrue from receiving correct and accurate information at the point of referral review. GPs and school staff advised that the system needs to guide them through the referral process and advise on alternative sources of help; the current processes are simply not fit for purpose and often cause distress to children and families.

Another key benefit of a standardised referral system is the ability to automatically collect data for onward reporting to national bodies (e.g. waiting times to NHS England). This automatic data collection would further enable benchmarking of CAMHS referral processes widely across and within Trusts in the UK. This monitoring of service performance in turn can provide a means for responding to problems quickly, as well as targeting support to areas where there are clear challenges.

RESEARCH QUESTION/AIM(S) The overarching aim is to improve the CAMHS referral process for CYP, their families and carers, as well as for health, education and CAMHS professionals so that CYP receive the help they need as quickly as possible.

Research questions:

1. Using the findings from EN-CAMHS 1 and stakeholder consultation, can the project team develop a set of national standards for digital CAMHS referral processes?
2. Can the project team translate the prioritised features from EN-CAMHS 1 of a digitally-led, intelligent CAMHS referral process into a usable, acceptable and widely accessible platform that is nationally standardised, locally adaptable and sustainable?
3. Can the project team address concerns about digital exclusion and other identified health inequalities through the newly developed CAMHS referral mechanisms?
4. How do referrers, including GPs, school staff and children/young people/families perceive the usability and acceptability of the digital tool?
5. How do referrers use and engage with the tool?
6. How do rates of successful referrals with the tool compare to traditional modes of referral?

Objectives

1. To develop national standards for digital referrals into CAMHS that have sufficient flexibility to support the diversity of CAMHS configurations locally and regionally (WP1).
2. To co-develop with key stakeholders a standards-compliant digital CAMHS referral tool that maximises the use of digital technologies to support inclusion (e.g. translation support, text to speech, culturally-relevant service information and imagery) (WP2).
3. To implement, test and refine the newly developed standards and digital tool in 5-8 CAMHS providers (WP3), with CAMH sites purposively selected for diverse contextual characteristics.
4. To develop a blueprint for implementation of the new referral process at CAMHS.
5. To develop a robust sustainability plan for standards-compliant CAMHS referral processes so that the platforms developed through the funding remain relevant, usable and useful beyond the lifetime of this grant funding (WP4).

Outcome To the project team's knowledge, this is the first study designed specifically to develop a solution to the challenge of rejected/inappropriate CAMHS referrals. Through extensive consultation with all key stakeholders on the referral process throughout EN-CAMHS 1, the project team are now positioned to build a solution to the problems of referral that addresses the needs of all types of referrers, including notably young people and their families. The project team's broad network of collaborators and partners on the project will support widespread dissemination of the work. The project team's partner MQ will work closely with the project team throughout the project to ensure dissemination, outputs and impact are maximised for the benefit of young people who require mental health support. As in EN-CAMHS 1, the project team shall leverage the project team's extensive mental health networks to influence and support policy change to bring benefit to CYP and their families through an enhanced referral process. The project team will aim to share findings as soon as possible and tailor these to the audience. The project team shall do this through ongoing updates through social media channels and those of the project team's partners (critically, MQ) and through ongoing presentations, conferences, seminars and informal events across the full lifetime of the project. MQ is the dissemination partner and the project team shall hold events with stakeholders throughout the project as part of the parallel work on implementation.

The project has the potential for far-reaching and sustained impact. Specifically, the project team anticipate and will aim for the following effects:

* Reduced proportion of inappropriate referrals to CAMHS.
* Greater proportion of successful referrals.
* Reduced clinical costs for use by CAMHS assessing CYP and families in need.
* Reduced waiting times for first appointments.
* Flattening of recent increases in referral rates.
* Improved quality of referrals and information therein.
* Reduction in length of initial referral meetings.
* Fewer delays in decision-making.
* Improved information about alternative services or self-help.
* With swifter processes, it will help reduce the number of young people who get to assessment stages and then get rejected for becoming eligible for adult services [9].
* Improved patient experience through transparency of progress during referral.
* Potentially more time made available for face to face appointments when needed due to more efficient and complete referral process.
* In services where dedicated time to discuss referrals are not routine, greater availability can be carved out for direct contact (phone, email) to prevent inappropriate and rejected referrals, and to ensure those CYP who need be seen do so. This remains an essential clinical activity to ensure patient safety. It would reduce the need for lengthy, and weekly referral meetings freeing up resource internally.
* Having the necessary sources of information and complete investigations prior to the initial assessment will improve throughput and waiting times within the CAMHS system leading to increased patient and clinician satisfaction and earlier interventions/diagnosis as appropriate Clinicians would be freed up from chasing further information to supplement their assessment and formulation and this will improve efficiency and release their time for clinical duties.
* The project team shall facilitate NHS England's ability to benchmark and monitor referrals into CAMHS and the information from the digital referrals process will also aid ICBs to commission services best suited to support local need.
* The project team shall influence policy and practice through direct contact with NHS partners and governments and by feeding information about referral over time and different regions. Many of the project team and collaborators are influencers at national and regional policy level (e.g. Abel; Chitsabesan; Ranote; Jiva). The project team shall also input directly to professional groups (e.g. Faculty of Child and Adolescent Psychiatry).

ELIGIBILITY:
Inclusion Criteria

Participants recruited will:

1. Have capacity to consent.
2. Be 16 years or over.
3. Be a CAMHS stakeholder who has had experience with the CAMHS referral process:

   CAMHS Staff: we will include any staff who currently work in CAMHS services Collaborators: We will include collaborators who have direct experience of the current referral process for CAMHS Children and Young People (CYP): We will be recruiting CYP who have been referred to CAMHS regardless of whether they were accepted into the service or not. CYP will be aged 16-30, and will have experience of the CAMHS referral process in the past 5 years.

   Key referrers: We would ask that these individuals have had experience referring CYP to CAMHS, regardless of how many times.

   Parents/carers: we will ask parents/carers who have experience of their child or a child in their care having been referred to CAMHS, regardless of the outcome of the referral. CAMHS Commissioners: We will ask Commissioners who understand the current CAMHS referral processes locally or nationally, and who are involved in the funding process Mental Health Leads: We will invite people with a strategic overview of the CAMHS referral process locally or nationally to share their experiences of the referral process.
4. Be proficient in English (or a supported language of the translated referral process).

Exclusion Criteria

1. People unable to speak and understand written English at a relatively high level.
2. People without good internet access to take part in the online focus groups.
3. People who have not had experience with the CAMHS referral process.
4. People who lack the capacity to consent.
5. Young people who are currently accessing CAMHS for support.

Regarding any level of illness/disability:

We feel it is up to the young person to make this decision during the consent process, and we could not make that decision for them. We will inform participants during the consent process (i.e. in the PIS and subsequent discussions) that there may be discussion which they could find upsetting, and we have a distress protocol in place for if anyone needs additional support, but that this should be considered when agreeing to take part in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Professionals, young people and parents/carers who have experience of the CAMHS referral process.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 2 months
  If the referral tool improves the experience of referral process, using data collected during focus groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
It is not required for IPD to be shared as part of this study.

REFERENCES:
- [Background] 1. Department of Health and Social Care (2023). URL: https://healthmedia.blog.gov.uk/2023/06/09/how-we-are-supporting-mental-health-services-in-england/ (accessed 25 July 2023)
- [Background] 2. Children's Mental Health Services 2021/22 (2023). Children's Commissioner. URL: https://assets.childrenscommissioner.gov.uk/wpuploads/2023/03/Childrens-Mental-Health-Services-2021-2022-2.pdf (accessed 25 July 2023)
- [Background] 3. Korkodilos M. The mental health of children and young people in England. London: Public Health England. 2016. https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_d ata/file/575632/Mental_health_of_children_in_England.pdf (accessed 25 July 2023)
- [Background] 4. Newlove-Delgado, T., Williams, T., Robertson, K., McManus, S., Sadler, K., Vizard, T., Cartwright, C., Mathews, F., Norman, S., Marcheselli, F. and Ford, T., 2021. Mental Health of Children and Young People in England 2021-wave 2 follow up to the 2017 survey. https://openaccess.city.ac.uk/id/eprint/28718/1/
- [Background] 5. McNicholas, F., Kelleher, I., Hedderman, E., Lynch, F., Healy, E., Thornton, T., Barry, E., Kelly, L., McDonald, J., Holmes, K. and Kavanagh, G., 2021. Referral patterns for specialist child and adolescent mental health services in the Republic of Ireland during the COVID-19 pandemic compared with 2019 and 2018. BJPsych open, 7(3), p.e91. https://doi.org/10.1192/bjo.2021.48
- [Background] 6. Grant, C., Blackburn, R., Harding, D., Golden, S., Toth, K., Scott, S., Ford, T. and Downs, J., 2023. Impact of counselling provision in primary schools on child and adolescent mental health service referral rates: a longitudinal observational cohort study. Child and Adolescent Mental Health, 28(2), pp.212-220. https://doi.org/10.1111/camh.12519
- [Background] 7. YoungMinds (2022). URL: https://www.youngminds.org.uk/about-us/media-centre/press-releases/mental-health-waiting-times-harming-young-people/ (accessed 25 June 2023)
- [Background] 8. Iskra, W., Deane, F.P., Wahlin, T. and Davis, E.L., 2018. Parental perceptions of barriers to mental health services for young people. Early intervention in psychiatry, 12(2), pp.125-134. https://doi.org/10.1111/eip.12281
- [Background] 9. Hansen, A.S., Telléus, G.K., Mohr-Jensen, C. and Lauritsen, M.B., 2021. Parent-perceived barriers to accessing services for their child's mental health problems. Child and Adolescent Psychiatry and Mental Health, 15, pp.1-11. https://doi.org/10.1186/s13034-021-00357-7
- [Background] 10. Scottish Government (2018). URL: https://www.gov.scot/binaries/content/documents/govscot/publications/research-and-analysis/2018/06/rejected-referrals-child-adolescent-mental-health-services-camhs-qualitative-quantitative/documents/00537523-pdf/00537523-pdf/govscot%3Adocument/00537523.pdf (accesses 26 July 2023)
- [Background] 11. Crouch, L., Reardon, T., Farrington, A., Glover, F. and Creswell, C., 2019. "Just keep pushing": Parents' experiences of accessing child and adolescent mental health services for child anxiety problems. Child: Care, Health and Development, 45(4), pp.491-499. https://doi.org/10.1111/cch.12672
- [Background] 12. Smith, J., Kyle, R.G., Daniel, B. and Hubbard, G., 2018. Patterns of referral and waiting times for specialist Child and Adolescent Mental Health Services. Child and Adolescent Mental Health, 23(1), pp.41-49. https://doi.org/10.1111/camh.12207
- [Background] 13. Royal College of Paediatrics and Child Health. URL: https://www.rcpch.ac.uk/news-events/news/school-referrals-mental-health-treatment-rise-third#:~:text=RCPCH's%20Dr%20Max%20Davie%20responds,in%20the%20last%20three%20years (accessed 26 July 2023)
- [Background] 14. Education and Health Select Committees. URL: https://publications.parliament.uk/pa/cm201617/cmselect/cmhealth/849/849.pdf (accessed 26 July 2023)
- [Background] 15. Lambert, A.K., Doherty, A.J., Wilson, N., Chauhan, U. and Mahadevan, D., 2020. GP perceptions of community-based children's mental health services in Pennine Lancashire: a qualitative study. BJGP open, 4(4). https://doi.org/10.3399/bjgpopen20X101075
- [Background] 16. Hinrichs, S., Owens, M., Dunn, V. and Goodyer, I., 2012. General practitioner experience and perception of Child and Adolescent Mental Health Services (CAMHS) care pathways: a multimethod research study. BMJ open, 2(6), p.e001573. http://dx.doi.org/10.1136/bmjopen-2012-001573
- [Background] 17. Evans, N. and Huws-Thomas, M., 2020. Case note review of community mental health services for children and young people in a UK rural location. The Journal of Mental Health Training, Education and Practice, 15(3), pp.171-179. https://doi.org/10.1108/JMHTEP-10-2019-0055
- [Background] 18. Abel, K.M., Whelan, P., Carter, L., Elvins, R., Edbrooke-Childs, J., Bunting, S., Stockton-Powdrell, C., Tranter, H., Gutridge, K., Hassan, L. (2022). Enhancing CAMHS Referrals ("ENCAMHS 1"). NIHR131379.
- [Background] 19. NHS Benchmarking Network (2019). URL: https://www.nhsbenchmarking.nhs.uk/news/2019-child-and-adolescent-mental-health-services-project-results-published (accessed 25 July 2023)
- [Background] 20. Hansen, A.S., Christoffersen, C.H., Telléus, G.K. and Lauritsen, M.B., 2021. Referral patterns to outpatient child and adolescent mental health services and factors associated with referrals being rejected. A cross-sectional observational study. BMC Health Services Research, 21, pp.1- 12. https://doi.org/10.1186/s12913-021-07114-8
- [Background] 21. Patalay, P. and Fitzsimons, E., 2017. Mental ill-health among children of the new century: trends across childhood with a focus on age 14. London: Centre for Longitudinal Studies, pp.1-6. URL: http://www.cls.ioe.ac.uk/shared/get-file.ashx?itemtype=document&id=3338 (accessed 25 July 2023)
- [Background] 22. Frith E. Access and waiting times in children and young people's mental health services. (2017). URL: https://epi.org.uk/wp- content/uploads/2018/01/EPI_Access-and-waiting-times_.pdf (accessed 25 July 2023)
- [Background] 23. Frith, E., 2016. Progress and challenges in the transformation of children and young people's mental health care. Education Policy Institute, London. URL:https://epi.org.uk/wp- content/uploads/2018/01/progress-and-challenges.pdf (accessed 25 July 2023)
- [Background] 24. Scottish Government (2018). URL: https://www.gov.scot/publications/rejected-referrals-child- adolescent-mental-health-services-camhs-qualitative-quantitative/pages/3/ (accessed 25 July 2023)
- [Background] 25. Care Quality Commission (CQC) (2018). URL: https://www.cqc.org.uk/publications/themed-work/are-we-listening-review-children-young-peoples-mental-health-services (accessed 25 July 2023)
- [Background] 26. Fazel, M., Rocks, S., Glogowska, M., Stepney, M. and Tsiachristas, A., 2021. How does reorganisation in child and adolescent mental health services affect access to services? An observational study of two services in England. PloS one, 16(5), p.e0250691. https://doi.org/10.1371/journal.pone.0250691
- [Background] 27. Rocks, S., Glogowska, M., Stepney, M., Tsiachristas, A. and Fazel, M., 2020. Introducing a single point of access (SPA) to child and adolescent mental health services in England: a mixed-methods observational study. BMC health services research, 20, pp.1-11. https://doi.org/10.1186/s12913-020-05463-4
- [Background] 28. The Children and Young People's Mental Health Taskforce. (2015). URL: https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/414024/Childrens_Mental_Health.pdf (accessed 25 July 2023)
- [Background] 29. The MoSCow Method (2023). URL: https://www.mindtools.com/a4xmovt/the-moscow-method (accessed 25 June 2023)
- [Background] 30. System usability scale. URL: https://www.usability.gov/how-to-and-tools/methods/system- usability-scale.html (accessed 14 March 2023)
- [Background] 31. Web Content Accessibility Guidelines (WCAG) 2.2. URL: https://www.w3.org/TR/WCAG22/ (accessed 20 May 2024)
- [Background] 32. Greenhalgh, T., Maylor, H., Shaw, S., Wherton, J., Papoutsi, C., Betton, V., Nelissen, N., Gremyr, A., Rushforth, A., Koshkouei, M. and Taylor, J., 2020. The NASSS-CAT tools for understanding, guiding, monitoring, and researching technology implementation projects in health and social care: protocol for an evaluation study in real-world settings. JMIR research protocols, 9(5), p.e16861. https://doi.org/10.2196/16861
- [Background] 33. Murray, E., Treweek, S., Pope, C., MacFarlane, A., Ballini, L., Dowrick, C., Finch, T., Kennedy, A., Mair, F., O'Donnell, C. and Ong, B.N., 2010. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC medicine, 8, pp.1-11. https://doi.org/10.1186/1741-7015-8-63
- [Background] 34. NHS BaRS standard (2023). URL: https://digital.nhs.uk/services/booking-and-referral-standard (accessed 25 June 2023)
- [Background] 35. NHS App (2023. URL: https://www.nhs.uk/nhs-app/about-the-nhs-app/ (accessed 25 June 2023)
- [Background] 36. Greenhalgh, T., Wherton, J., Papoutsi, C., Lynch, J., Hughes, G., Hinder, S., Fahy, N., Procter, R. and Shaw, S., 2017. Beyond adoption: a new framework for theorizing and evaluating nonadoption, abandonment, and challenges to the scale-up, spread, and sustainability of health and care technologies. Journal of medical Internet research, 19(11), p.e8775. https://doi.org/10.2196/jmir.8775
- [Background] 37. Agile delivery (2023). URL: https://www.gov.uk/service-manual/agile-delivery (accessed 25 June 2023)
- [Background] 38. How the discovery phase works (2021). URL: https://www.gov.uk/service-manual/agile-delivery/how-the-discovery-phase-works (accessed 25 June 2023)
- [Background] 39. How the alpha phase works (2019). URL: https://www.gov.uk/service-manual/agile-delivery/how-the-alpha-phase-works (accessed 25 June 2023)
- [Background] 40. How the beta phase works (2021). URL: https://www.gov.uk/service-manual/agile-delivery/how-the-beta-phase-works (accessed 25 June 2023)
- [Background] 41. How the live phase works (2019). URL: https://www.gov.uk/service-manual/agile-delivery/how-the-live-phase-works (accessed 25 June 2023)
- [Background] 42. Amused Framework : Miller S, Ainsworth B, Yardley L, Milton A, Weal M, Smith P, Morrison L A Framework for Analyzing and Measuring Usage and Engagement Data (AMUsED) in Digital Interventions: Viewpoint J Med Internet Res 2019;21(2):e10966. https://doi.org/10.2196/10966
- [Background] 43. Ritchie, J. and Spencer, L., 2002. Qualitative data analysis for applied policy research. In Analyzing qualitative data (pp. 173-194). Routledge.
- [Background] 44. Ritchie, J., Lewis, J., Nicholls, C.M. and Ormston, R. eds., 2013. Qualitative research practice: A guide for social science students and researchers. sage.
- [Background] 45. Nvivo 11 (n.d.). URL: https://help - nv11.qsrinternational.com/desktop/concepts/about_framework_matrices.htm (accessed 25 June 2023).
- See also: NIHR Funding Awards — https://fundingawards.nihr.ac.uk/award/NIHR158809
- See also: GM.Digital Research Unit website for project updates — https://camhs.digital/

DOCUMENTS (2):
  • Study Protocol: Study_Protocol (2025-10-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT07399106/Prot_000.pdf
  • Informed Consent Form (2025-10-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT07399106/ICF_001.pdf